CLINICAL TRIAL: NCT00702715
Title: A Multi-center, Parallel-group, Comparative Trial Evaluating the Efficacy, Pharmacokinetics and Safety of 4.0 mg/kg Sugammadex Administered at 1-2 PTC in Subjects With Normal or Severely Impaired Renal Function
Brief Title: Comparison of 4.0 mg/kg Sugammadex at 1-2 Post Tetanic Counts (PTC) in Renal or Control Patients (19.4.328)(P05769)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05769; 19.4.328
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2011-04-11 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants with severe renal impairment (Experimental): Participants with severe renal impairment will receive a single bolus dose of 4.0 mg.kg-1 sugammadex at a target depth of blockade of 1-2 PTC. Severe renal impairment was defined as creatinine clearance <30mL/min.
  Interventions: Drug: sugammadex
- Participants with normal renal function (Active Comparator): Participants with normal renal impairment will receive a single bolus dose of 4.0 mg.kg-1 sugammadex at a target depth of blockade of 1-2 PTC. Normal renal function was defined as creatinine clearance >=80mL/min.
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex — Each subject will receive an
  intravenous (i.v.) single bolus dose of 0.6 mg.kg-1 rocuronium. After
  this dose, maintenance doses of 0.1 - 0.2 mg.kg-1
  rocuronium may be given. In case of maintenance dosing, the target depth of
  neuromuscular blockade has to be maintained at 1-2 post-tetanic counts (PTC). After the last dose of rocuronium has been administered, the subject will receive a single bolus dose of 4.0 mg.kg-1 sugammadex at a target depth of blockade of 1-2 PTC.
  Other Names: Org 25959

SUMMARY:
The current trial was designed to investigate the effects of 4.0 mg.kg-1 of sugammadex on efficacy, safety and pharmacokinetics in subjects with severe renal impairment in comparison to subjects with normal renal function.

DETAILED DESCRIPTION:
The results of previous trials showed that the safety profile of sugammadex

observed in subjects with impaired renal function are not appreciably different from subjects with normal renal function. Reoccurrence of neuromuscular blockade was not observed, and sugammadex was safe and generally well tolerated in subjects with severe renal impairment. In a previous trial, subjects (n=15) with severe renal impairment received a dose of 2.0 mg.kg-1 of sugammadex. The effects of the other proposed recommended dose for routine reversal, 4.0 mg.kg-1, on efficacy, safety and pharmacokinetics had not been studied thus far in subjects with severe renal impairment. The objectives of this trial were to assess equivalence with respect to the efficacy of sugammadex in subjects with normal renal function or severe renal impairment, to evaluate the safety of sugammadex in these subject groups and to compare the pharmacokinetic profiles.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* ASA class 1-3
* Creatinine clearance (CLcr) < 30 mL/min and no anticipated clinical

indication for high flux hemodialysis during first 24 hours after

sugammadex administration (for renally impaired group) or CLcr >= 80

mL/min (for control group)

-Scheduled for a surgical procedure under general anesthesia with propofol

requiring neuromuscular relaxation with the use of rocuronium

* Scheduled for a surgical procedure in supine position
* Written informed consent

Exclusion Criteria:

- Subjects known or suspected to have neuromuscular disorders impairing

neuromuscular blockade and/or significant hepatic dysfunction

* Subjects scheduled for renal transplant surgery
* Subjects known or suspected to have a (family) history of malignant

hyperthermia

-Subjects known or suspected to have an allergy to narcotics, muscle

relaxants or other medication used during general anesthesia

* Subjects receiving fusidic acid, toremifene and/or flucloxacillin
* Subjects who have already participated in a sugammadex trial
* Subjects who have participated in another clinical trial, not pre-approved

by the sponsor, within 30 days of entering into 19.4.328 (P05769)

* Female subjects who are pregnant
* Female subjects who are breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-09-24 (Actual); Primary Completion 2010-03-15 (Actual); Study Completion 2010-03-15 (Actual)

REFERENCES:
- [Result] Panhuizen IF, Gold SJ, Buerkle C, Snoeck MM, Harper NJ, Kaspers MJ, van den Heuvel MW, Hollmann MW. Efficacy, safety and pharmacokinetics of sugammadex 4 mg kg-1 for reversal of deep neuromuscular blockade in patients with severe renal impairment. Br J Anaesth. 2015 May;114(5):777-84. doi: 10.1093/bja/aet586. Epub 2015 Mar 31. PMID 25829395

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Severe Renal Impairment: Participants with severe renal impairment will receive a single bolus dose of 4.0 mg.kg-1 sugammadex at a target depth of blockade of 1-2 post-tetanic counts (PTC). Severe renal impairment was defined as creatinine clearance <30mL/min.
Period: Overall Study
Arm/Group | Participants With Severe Renal Impairment | Participants With Normal Renal Function
Started | 35 | 33 (One subject was enrolled but did not start study)
Completed | 34 | 33
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Severe Renal Impairment | Participants With Normal Renal Function | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (16) | 45 (15) | 51 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery of the T4/T1 Ratio to 0.9.
Description: Neuromuscular functioning was monitored by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. Nerve stimulation continued until the ratio of the magnitude of the fourth twitch (T4) to first twitch (T1) reached at least 0.9. The greater the T4/T1 ratio the greater the recovery from neuromuscular blockade, with a value of 1.0 representing full recovery.
Time Frame: start of administration of sugammadex to recovery from neuromuscular blockade
Population: Analysis performed using the Intent-to-Treat (ITT) Population, which consisted of all treated subjects who had at least one efficacy measurement.
Measure: Geometric Mean (95% Confidence Interval); unit: seconds
Arm/Group | Participants With Severe Renal Impairment | Participants With Normal Renal Function
Number analyzed (Participants) | 35 | 32
seconds | 205 [169 to 248] | 112 [92 to 138]
Statistical Analysis 1: Comparison: Participants With Severe Renal Impairment vs Participants With Normal Renal Function; Test type: Non-Inferiority or Equivalence — The 95% confidence interval for the estimated median treatment difference in recovery time must have fallen entirely within the pre-specified interval between -60 sec to +60 sec in order to claim equivalence; Hodges-Lehmann and Moses; Median Difference (Final Values) = 78.0, 95% CI 2-sided [36.0 to 143.0] — Estimated median treatment difference (severe renal impairment minus normal renal function) in recovery time (seconds)

2. Secondary Outcome: Time to Recovery of the T4/T1 Ratio to 0.8
Description: as for outcome 1
Time Frame: start of administration of sugammadex to recovery from neuromuscular blockade
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: seconds
Arm/Group | Participants With Severe Renal Impairment | Participants With Normal Renal Function
Number analyzed (Participants) | 35 | 32
seconds | 169 [141 to 203] | 90 [76 to 107]
Statistical Analysis 1: Comparison: Participants With Severe Renal Impairment vs Participants With Normal Renal Function; Test type: Non-Inferiority or Equivalence — For the secondary endpoint no equivalence margin was specified (i.e., no formal null-hypothesis was specified); the median difference and associated 95% CI were to further characterize the efficacy of severe renal impaired subjects and controls; Hodges-Lehmann and Moses; Median Difference (Final Values) = 68.0, 95% CI 2-sided [36.0 to 120.0] — Estimated median treatment difference (severe renal impairment minus normal renal function) in recovery time (seconds)

3. Secondary Outcome: Time to Recovery of T4/T1 Ratio to 0.7
Description: as for outcome 1
Time Frame: start of administration of sugammadex to recovery from neuromuscular blockade
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: seconds
Arm/Group | Participants With Severe Renal Impairment | Participants With Normal Renal Function
Number analyzed (Participants) | 35 | 32
seconds | 144 [120 to 172] | 79 [67 to 92]
Statistical Analysis 1: Comparison: Participants With Severe Renal Impairment vs Participants With Normal Renal Function; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Hodges-Lehmann and Moses; Median Difference (Final Values) = 60.0, 95% CI 2-sided [31.0 to 103.0] — Estimated median treatment difference (severe renal impairment minus normal renal function) in recovery time (seconds)

ADVERSE EVENTS:
Arm/Group | Participants With Severe Renal Impairment | Participants With Normal Renal Function
Serious Adverse Events (participants affected / at risk) | 9/35 | 3/33
Other Adverse Events (participants affected / at risk) | 14/35 | 17/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Severe Renal Impairment (N=35) | Participants With Normal Renal Function (N=33)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Thrombophlebitis septic (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Narcotic intoxication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Severe Renal Impairment (N=35) | Participants With Normal Renal Function (N=33)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 9 (9) | 11 (13)
Neutrophil count increased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All published results will be based on validated data released by the sponsor and must include one sponsor author. There may be one author from each investigational site, provided that the criteria for authorship are met. In case the proposed publication contains reference to an invention owned by sponsor or to which sponsor otherwise has rights, the sponsor may request a reasonable suspension of the publication in order to be able to file a patent application protecting such invention.